CLINICAL TRIAL: NCT00002972
Title: Phase II Study on TAXOL in Bronchioalveolar Carcinoma
Brief Title: Paclitaxel in Treating Patients With Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-08956; EORTC-08956
Record Dates: First submitted 1999-11-01; First posted 2003-04-17 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients who have unresectable stage IIIB, stage IV or recurrent lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the therapeutic activity of paclitaxel in patients with bronchoalveolar carcinoma (BAC).
* Assess the duration of response in patients presenting with an objective response.
* Characterize the acute side effects of paclitaxel in patients with BAC.
* Assess the role of some biological parameters in the natural history and the response to therapy of BAC; evaluate the expression of Ki67, p53, and K-ras mutation.

OUTLINE: This is an open label, nonrandomized, multicenter study.

Paclitaxel is administered every 3 weeks as a 3 hour continuous infusion in dextrose or normal saline. Patients are treated for a minimum of 2 cycles unless serious toxicity or complication occur.

Disease is assessed every 6 weeks until documented progression; treatment side effects are assessed separately for each cycle of therapy. Treatment is given up to a maximum of 6 cycles of therapy or until disease progression, unacceptable toxicity, or patient refusal occurs.

PROJECTED ACCRUAL: 16 or 25 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven bronchoalveolar carcinoma (BAC) based on these criteria:

  * Absence of primary adenocarcinoma elsewhere
  * Absence of a demonstrable central bronchogenic origin
  * A peripheral location in the lung parenchyma
  * Intact interstitial framework of the lung
  * A histological appearance setting it apart from other tumors, with a characteristic pattern of growth: cuboidal or cylindrical cells lining up the alveolar septa with preservation of basic pulmonary architecture
* Must be unresectable Stage IIIB, IV, or recurrent BAC
* Evidence of multinodular lesions involving the lungs bilaterally or unilaterally (in the latter the lesions must involve more than one lobe)
* At least one target lesion bidimensionally measurable that has not undergone prior irradiation
* No CNS disease

PATIENT CHARACTERISTICS:

Age:

* 18 to 75 (inclusive)

Performance status:

* ECOG 0-2

Life expectancy:

* Greater than 3 months

Hematopoietic:

* ANC at least 1,500/mm^3

Hepatic:

* Bilirubin less than 2 times upper limit of normal
* SGOT, SGPT, and alkaline phosphatase less than 2 times upper limit of normal

Renal:

* Creatinine less than 1.5 times upper limit of normal

Cardiovascular:

* No history of ischemic or congestive heart disease
* No arrhythmia requiring chronic cardiopulmonary medications
* No history of clinically or electrographically documented myocardial infarction

Other:

* No preexisting motor or other serious sensory neurotoxicity
* No active or prior second primary cancer except basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No clinical evidence of uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test 72 hours prior to start of study medication
* Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since radiotherapy
* Must have at least one bidimensional lesion outside the irradiated fields

Surgery:

* Fully recovered from any prior major surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1997-01; Primary Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Scagliotti, MD, PhD, Study Chair — Azienda Ospedale S. Luigi at University of Torino
Locations (5):
- Centre Hospitalier Regional de la Citadelle, Liege (Luik), Belgium
- University Thomayers' Hospital, Krhanice, Czechia
- Universitaetsklinik und Strahlenklinik - Essen, Essen, Germany
- Azienda Ospedale S. Luigi - Universita Di Torino, Orbassano, (Torino), Italy
- Vrije Universiteit Medisch Centrum, Amsterdam, Netherlands

REFERENCES:
- [Result] Scagliotti GV, Smit E, Bosquee L, O'Brien M, Ardizzoni A, Zatloukal P, Eberhardt W, Smid-Geirnaerdt M, de Bruin HG, Dussenne S, Legrand C, Giaccone G; European Organisation for Research and Treatment of Cancer (EORTC) Lung Cancer Group (LCG). A phase II study of paclitaxel in advanced bronchioloalveolar carcinoma (EORTC trial 08956). Lung Cancer. 2005 Oct;50(1):91-6. doi: 10.1016/j.lungcan.2005.05.012. PMID 16019107